CLINICAL TRIAL: NCT03980197
Title: Strategy to Prevent Transmission of Multidrug-resistant Gram-negative Organisms in ICU - Evaluation of Effect of Active Surveillance Test
Brief Title: Strategy to Prevent Transmission of Multidrug-resistant Gram-negative Organisms in ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sung-Han Kim (Other)
Responsible Party: Sponsor-Investigator, Sung-Han Kim, Princiapl investigator, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2019-0274
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Antibiotic Resistant Infection
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Active surveillance test and preemptive isolation is performed. If MDRO is isolated in surveillance test, contact precaution is needed.
  Interventions: Other: Active surveillance and preemptive isolation
- Control (Active Comparator): No active surveillance test and preemptive isolation performed. Only standard precaution is needed, and if clinical isolates reveals MDRO, start contact precaution.
  Interventions: Other: Control

INTERVENTIONS:
Other: Active surveillance and preemptive isolation — Active surveillance test and preemptive isolation is performed. If MDRO is isolated in surveillance test, contact precaution is needed.
  Arms: Intervention
Other: Control — No active surveillance and preemptive isolation. If clinical isolates are positive for MDRGNB, start contact precaution
  Arms: Control

SUMMARY:
1. Objective of study The purpose of this study was to investigate whether the active surveillance and preemptive isolation of multidrug-resistant Gram-negative bacteria in the intensive care unit affected the reduction of the rate of acquisition of multidrug- resistant Gram-negative bacteria (MDRGNB).
2. Background Treatment option for MDRGNB (Carbapenem-resistant P. aeruginosa, Carbapenem-resistant A. baumannii, Carbapenem-resistant Enterobacteriaceae) is limited. Development of infection due to MDRGNB is common in ICU. Strategy to prevent transmission of MDRGNB is needed, and there is two approaches; First, antimicrobial stewardship program, and second, infection control strategy.The investigators aimed to figure out the role of active surveillance test and preemptive isolation of MDRGNB in reduction of acquisition rate of MDRGNB.
3. Methods Pragmatic cluster randomized, crossover, controlled trial During first period (6 months), intervention group (randomized 3 ICUs) perform daily chlorhexidine bathing, active surveillance test and preemptive isolation and contact precaution. Control group (randomized 3 ICUs) perform standard precaution with daily chlorhexidine bathing, and start contact precaution when clinical isolates reveals MDRGNB.

After 1 month washout period, intervention group and control group cross over for next 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Enroll all patients who admit to the ICUs during the study period

Exclusion Criteria:

* Patients who discharge within 2 days after admission to ICUs

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2500 (Estimated)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
The number of patients who acquired MDRGNB in ICU per 1000 patient-days | through study completion, an average 6 months
  The number of patients who acquired MDRGNB in ICU per 1000 patient-days

SECONDARY OUTCOMES:
Rate of bloodstream infection due to MDRGNB | through study completion, an average 6 months
  Rate of bloodstream infection due to MDRGNB
Hand hygiene compliance rates (%) of healthcare workers | through study completion, an average 1 year
  number of Hand hygiene compliance/number of opportunicities for hand hygiene of healthcare workers *100
Days of ICU stay | through study completion, an average 6 months
  Days of ICU stay
28-day mortality rate | 28-days
  28-day mortality rate

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung J, Park JH, Yang H, Lim YJ, Kim EO, Lim CM, Kim MN, Jo MW, Yun SC, Kim SH. Active surveillance testing to reduce transmission of carbapenem-resistant, gram-negative bacteria in intensive care units: a pragmatic, randomized cross-over trial. Antimicrob Resist Infect Control. 2023 Mar 3;12(1):16. doi: 10.1186/s13756-023-01222-2. PMID 36869371